CLINICAL TRIAL: NCT00066144
Title: Black Cohosh and Red Clover Efficacy for the Relief of Menopausal Symptoms
Brief Title: Use of Black Cohosh and Red Clover for the Relief of Menopausal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Collaborators: Office of Dietary Supplements (ODS) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P50AT000155 (NIH)
Record Dates: First submitted 2003-08-04; First posted 2003-08-05 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Hot Flashes; Menopause
Keywords: menopause; hot flashes; red clover; black cohosh; sexual dysfunction
MeSH Terms: conditions — Hot Flashes; Sexual Dysfunction, Physiological | interventions — black cohosh root extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cimicifuga racemosa
Drug: Trifolium pratense
Drug: Black cohosh
Drug: Red clover

SUMMARY:
This Phase II study, a follow-up to a Phase I trial in normal volunteers, will determine the efficacy of black cohosh and red clover for the relief of menopausal symptoms. It will also assess the safety of chronic dosing (1 year) by evaluating uterine (endometrial biopsies), breast (mammography), and hematology parameters (CBC and chemistry lab values) at baseline and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women with intact uterus
* Must be experiencing hot flashes
* No menstrual periods for at least 6 months and no longer than 3 years
* Non-smoker
* Must have intact uterus (no hysterectomy)

Exclusion Criteria:

* Contraindications for hormone replacement therapy
* Diabetes mellitus
* Pregnancy or breast-feeding
* Obese (BMI >35 excluded)
* History of endometrial hyperplasia/neoplasia/malignancy
* History of breast or reproductive cancer
* History of severe recurrent depression, or severe psychiatric disturbance
* History of stroke/CVA, severe varicose veins, sickle cell anemia, myocardial infarction (heart attack), or arrhythmia (rhythm disturbance of the heart)
* History of abnormal vaginal bleeding of unknown cause
* Untreated or uncontrolled high blood pressure/hypertension
* Use of any medication or supplement containing estrogen, progestin, SERM, St. John's Wort, bisphosphonates, or phytoestrogens
* History of hormone-associated migraines
* History of deep vein thrombosis (blood clots), thrombophlebitis, or thromboembolic disorders
* Participation in a clinical trial within 30 days
* Abnormal endometrial biopsy or mammogram
* Abnormal transvaginal ultrasound defined as >7mm thickness
* Vegan

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2003-04; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Geller, MD, Principal Investigator — Department of Obstetrics and Gynecology University of Illinois, Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Geller SE, Shulman LP, van Breemen RB, Banuvar S, Zhou Y, Epstein G, Hedayat S, Nikolic D, Krause EC, Piersen CE, Bolton JL, Pauli GF, Farnsworth NR. Safety and efficacy of black cohosh and red clover for the management of vasomotor symptoms: a randomized controlled trial. Menopause. 2009 Nov-Dec;16(6):1156-66. doi: 10.1097/gme.0b013e3181ace49b. PMID 19609225